CLINICAL TRIAL: NCT04082143
Title: CATER: Comprehensive Alveolar and Tooth Esthetic Replacement
Acronym: CATER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Sandra Al-Tarawneh, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0255
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Dental Implant Failure Nos
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: subjects will be randomized to one of two groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Implant with prophylactic allograft (Experimental): Implant placement will be performed with simultaneous placement of the allograft.
  Interventions: Device: Allograft mucosal enhancement with dental implant
- Implant without prophylactic allograft (Active Comparator): Implant placement will be performed without a graft
  Interventions: Device: No allograft mucosal enhancement at time of dental implant placement

INTERVENTIONS:
Device: Allograft mucosal enhancement with dental implant — implant placement with allograft mucosal enhancement
  Arms: Implant with prophylactic allograft
Device: No allograft mucosal enhancement at time of dental implant placement — implant placement without allograft mucosal enhancement
  Arms: Implant without prophylactic allograft

SUMMARY:
The purpose of this study is to prospectively evaluate whether including an allogeneic gum graft (PerioDerm*) during dental implant therapy improves implant health and appearance.

On the day of implant surgery, participating subjects will be randomized to either receive or not receive a supplemental gum graft along with the implant. Participating subjects will also be asked to complete a brief (about 15 questions) oral health questionnaire.

Participating subjects will return to the clinic about 8 weeks post surgery for digital crown impressions and again at 11-13 weeks after surgery for crown placement. Participating subjects will also return to clinic at 1 year after implant placement for implant evaluation. At this final study appointment, x-rays and a 3D intraoral scan will be obtained for the purpose of measuring alveolar volume. The health of the mucosa surrounding the implant and subject satisfaction will be assessed via bleeding upon probing and completion of a brief questionnaire, respectively.

DETAILED DESCRIPTION:
An alveolar ridge is the part of the jawbone which immediately surrounds and anchors the tooth socket ("alveolus"). Similar to any bone or muscle atrophying when not used, the alveolar ridge will shrink ("resorb") following tooth extraction. The volume of an alveolar ridge can be measured by both 3 Dimensional ("3D") intraoral scan and radiography, and is used clinically as a metric of oral health.

A dental implant is a medical-grade titanium screw placed into healed alveolar bone or a tooth socket following tooth extraction. It replaces the tooth root and supports the crown, or "dental cap"; an artificial tooth generally made with porcelain or surgical grade metals.

Implant success requires both sufficient bone alveolar volume and sufficient mucosal tissue to protect against biofilm-mediated inflammation, assure functional comfort and contribute to dental implant esthetics. Following dental implant placement, the alveolar ridge resorbs approximately 0.5 to 1.0 mm during the first year. Healed ridges are also often volumetrically deficient, losing up to 30% of their horizontal volume following tooth extraction.

To remedy this, peri-implant mucosal grafting has been proposed and is currently part of dental implant therapy. Both autogenous grafts (mucosal connective tissue from the roof of the patient's own mouth or "palate") and allogeneic grafts (collagen-rich grafts derived from a genetically non-identical human donor) are used for these purposes, but there is controversy regarding the effectiveness of supplemental graft use during implant treatment.

The purpose of this study is to prospectively evaluate whether including an allogeneic gum graft (PerioDerm*) during dental implant therapy improves implant health and appearance.

On the day of implant surgery, participating subjects will be randomized to either receive or not receive a supplemental gum allograft along with the implant. Participating subjects will also be asked to complete a brief (about 15 questions) oral health questionnaire.

Participating subjects will return to the clinic about 8 weeks post surgery for digital crown impressions and again at 11-13 weeks after surgery for crown placement. Participating subjects will also return to clinic about 1 year after implant placement for assessment of the implant evaluation. At this final study appointment, x-rays, a 3D intraoral scan and intraoral photographs of the implant will be obtained for the purpose of measuring alveolar volume. The health of the mucosa surrounding the implant and subject satisfaction will be measured via bleeding upon probing and completion of a brief questionnaire, respectively.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Willing and able to provide informed consent
* In need of one implant to replace a missing tooth
* At least 20 teeth in good repair and occlusion
* Sufficient bone volume for dental implant placement without required bone augmentation
* Site development (soft and/or bone tissue) performed at least 5 months before implant placement, when required

Exclusion Criteria:

* Current smoker
* Implant cannot be placed without bone graft
* Unable to pay for crown
* Untreated rampant caries and/or uncontrolled periodontitis
* Absence of adjacent (mesial and/or distal) natural tooth
* Uncontrolled diabetes
* Systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
* use of bisphosphonates
* History of radiation in the head and neck region
* Unable or unwilling to return for follow-up visits
* Unrealistic esthetic or functional demands
* Unlikely to be able to comply with study procedures
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-08-25 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Al-Tarawneh, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago College of Dentistry, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The target was to recruit a total of 40 participants (20 for each group) and up to 60 as a maximum. The number that was eventually enrolled in the study was 39.
Period: Overall Study
Arm/Group | Implant With Prophylactic Allograft | Implant Without Prophylactic Allograft
Started | 19 | 20
Completed | 19 | 18
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Implant With Prophylactic Allograft | Implant Without Prophylactic Allograft | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (3) | 53.1 (2) | 52.8 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 9 | 8 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Volume of Alveolar Ridge as Measured by 3D Intraoral Scanning
Description: Volume of the alveolar ridge (percentage change of the volume) as measured by 3D Intraoral scanning
Time Frame: 12 months post implant surgery
Measure: Mean (Standard Deviation); unit: percentage of volume change
Arm/Group | Implant With Prophylactic Allograft | Implant Without Prophylactic Allograft
Number analyzed (Participants) | 19 | 18
percentage of volume change | 15.5 (19) | 16.8 (62)

2. Secondary Outcome: Percentage of Implant Survival
Description: Implant survival at 12 months post implant surgery. Percentage of implants surviving after 12 months of placement
Time Frame: 12 months post implant surgery
Population: Two implants in the group (Implant without prophylactic allograft failed resulting in a 90% survival rate in that group and 95% overall survival rate for the study.
Measure: Number; unit: Percentage
Arm/Group | Implant With Prophylactic Allograft | Implant Without Prophylactic Allograft
Number analyzed (Participants) | 19 | 20
Percentage | 100 | 90

3. Secondary Outcome: Marginal Bone Levels (MBLs)
Description: Marginal bone levels (in millimeters) as measured by radiographic translucency. Bone levels between implant/abutment interface and crest of the bone were measured at time of implant placement and at 12 months later. The negative sign in the results below indicates that there was bone loss in both groups.
Time Frame: 12 months post implant surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Implant With Prophylactic Allograft | Implant Without Prophylactic Allograft
Number analyzed (Participants) | 19 | 18
mm | -0.17 (0.33) | -0.01 (0.11)

4. Secondary Outcome: Vertical Tissue Change as Measured by 3D Intraoral Scanning
Description: This measurement is for the vertical position of the gingival margin change based on superimposed 3D intraoral scans
Time Frame: 12 months post surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Implant With Prophylactic Allograft | Implant Without Prophylactic Allograft
Number analyzed (Participants) | 19 | 18
mm | 0.18 (0.27) | 0.16 (0.31)

5. Other Pre Specified Outcome: Patient Satisfaction
Description: Patient satisfaction with implant therapy as measured by the Oral Health Impact Profile
Time Frame: 12 months post implant surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Throughout the study from the time of enrollment until study closure which is marked by the one year follow up of the all participants who came back to that visit.
Description: All adverse events were monitored throughout the study period. The nature of standard routine implant placement procedure doesn't impose serious risk, and none of the participants experienced any adverse side effects.
Arm/Group | Implant With Prophylactic Allograft | Implant Without Prophylactic Allograft
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT04082143/Prot_SAP_001.pdf